CLINICAL TRIAL: NCT03409172
Title: Inflammatory and Metabolic Outcomes in Obese Women After 8 Weeks of High Intensity Interval Training and Moderate Intensity Continuous Training: a Randomized Controlled Pilot Study
Brief Title: Inflammatory and Metabolic Outcomes After Obese Woman Performed High Intensity Interval Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Vivian Marques Miguel Suen, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aerobic exercise and obesity
Record Dates: First submitted 2018-01-09; First posted 2018-01-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Obesity and Metabolic Syndrome
Keywords: High intensity interval training; Inflammation; Obesity; adipokines
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Inflammation

STUDY DESIGN:
Intervention Model Description: Three-arm parallel, Randomized-controlled study
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessors involved in data analysis will not be aware of the arm to which the participants were allocated (single-blinded masking)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (CTr) (Experimental): No counseling or nutritional therapy and no exercise
  Interventions: Other: CTR
- Moderate intensity continuous training (MICT) (Experimental): Follow-up during a period of 8 weeks of supervised ergometer-based moderate-intensity continuous training based on HRmax (MICT).
  MICT:
  * 3 sessions per week
  * intensity at 65-75% HRmax
  * time-effort per session: 50 min
  Interventions: Other: MICT
- High Intensity Interval Training (HIIT) (Experimental): Procedures: Follow-up during a period of 8 weeks of supervised ergometer-based high intensity interval training based on HRmax (HIIT).
  HIIT:
  * 3 sessions per week
  * 10 bouts of one minute at 90% HRmax interspersed by one minute at 40% HRmax
  * time-effort per session: 25 min
  Interventions: Other: HIIT

INTERVENTIONS:
Other: CTR — no counseling or nutritional therapy and no exercise
  Arms: Control group (CTr)
Other: MICT — no counseling or nutritional therapy. 8 weeks of individualized and supervised ergometer-based moderate continuous intensity training (MICT).
  Arms: Moderate intensity continuous training (MICT)
Other: HIIT — no counseling or nutritional therapy. 8 weeks of individualized and supervised ergometer-based high intensity interval training (HIIT)
  Arms: High Intensity Interval Training (HIIT)

SUMMARY:
The main purpose of this study is to compare the effects of high intensity interval training and moderate intensity continuous training on inflammatory profile and metabolic markers, after 8 weeks of intervention trial in obese women.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between (30-40 kg/m²)
* age between 25 and 41 years
* to be sedentary

Exclusion Criteria:

* type 1 or type 2 diabetes
* Hypertension
* pregnancy, Lactation
* having undergone bariatric surgery
* psychological disorders, epilepsy, sever neurological disorders
* participation in other moderate, vigorous exercise or nutrition intervention
* acute or chronic cardiovascular disease
* malignant disease
* kidney disease
* lung disease
* hyperthyroidism or hypothyroidism
* smoking any type of cigarette
* joint limitations
* electronic implants (defibrillator, pacemaker)

Ages: 25 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Inflammatory profile | 8 weeks (baseline to 8 week follow-up assessment)
  C-reactive protein (CRP) (mg/dL)
Inflammatory profile | 8 weeks (baseline to 8 week follow-up assessment)
  Interleukin 6 (IL-6) (ng/mL)
Inflammatory profile | 8 weeks (baseline to 8 week follow-up assessment)
  Interleukin 10 (IL-10) pg/mL, Interleukin-1B (IL-1B) pg/mL, Tumor Necrosis Factor (TNF)-α (pg/mL), Adiponectin (pg/mL), Monocyte chemoattractant protein 1 (MCP-1) (pg/mL), Leptin (pg/mL)

SECONDARY OUTCOMES:
Body Composition and Anthropometric profile | 8 weeks (baseline to 8 week follow-up assessment) ]
  Body weight (kg), Fat free mass (FFM) (kg), fat mass (FM) (kg)
Body Composition and Anthropometric profile | 8 weeks (baseline to 8 week follow-up assessment) ]
  Body Mass Index (BMI) (kg/m²)
Body Composition and Anthropometric profile | 8 weeks (baseline to 8 week follow-up assessment) ]
  Waist circumference (cm), hip circumference (cm)
Body Composition and Anthropometric profile | 8 weeks (baseline to 8 week follow-up assessment) ]
  Body Adiposity Index (BAI) and Waist-To-Hip Ratio (WHR)
Insulin sensitivity | 8 weeks (baseline to 8 week follow-up assessment) ]
  Insulin sensitivity was estimated using homeostasis model assessment index (HOMA)
Lipid profile | 8 weeks (baseline to 8 week follow-up assessment) ]
  Lipid profile was assessed by measuring levels of triglyceride (TG) (mg/dL), total cholesterol (CT) (mg/dL), high-density lipoprotein cholesterol (HDL-C) (mg/dL) and low-density lipoprotein cholesterol (LDL-C) (mg/dL)
Cardiorespiratory Fitness (CRF) | 8 weeks (baseline to 8 week follow-up assessment) ]
  CRF was assessed by measuring Peak Oxygen uptake (VO2peak) mL/kg/min
Blood Pressure (BP) | 8 weeks (baseline to 8 week follow-up assessment) ]
  Blood Pressure (mmHg) was assessed by measuring rest levels of Systolic blood pressure (SBP) and Diastolic blood pressure (DBP)
Resting Energy Expenditure (REE) | 8 weeks (baseline to 8 week follow-up assessment) ]
  Resting Energy Expenditure (kcal/day) was measured through indirect calorimetry with an open-circuit ventilated-hood system Substrate oxidation rate was calculated from VO2 (mL/min) and VCO2 (mL/min)
Substrate oxidation rate | 8 weeks (baseline to 8 week follow-up assessment) ]
  Substrate oxidation rate was calculated from VO2 (mL/min) and VCO2 (mL/min)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian M M SUEN, PhD, Study Director — fmrp usp

IPD SHARING:
Plan to Share IPD: No